CLINICAL TRIAL: NCT00027222
Title: The Early Treatment for Retinopathy of Prematurity Study (ETROP)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Purpose: Treatment
Other Study IDs: NEI-83
Record Dates: First submitted 2001-11-28; First posted 2001-10-29 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

INTERVENTIONS:
Procedure: retinal ablation

SUMMARY:
The goal of the Early Treatment for Retinopathy of Prematurity Study (ETROP) is to test the hypothesis that earlier treatment in carefully selected cases will result in an overall better visual outcome than treatment at the conventional CRYO-ROP threshold point in the disease.

DETAILED DESCRIPTION:
At age 5 1/2 years, the oldest age for which follow-up data are available, children with threshold ROP who were enrolled in the Cryotherapy for Retinopathy of Prematurity (CRYO-ROP) -- Outcome Study showed fewer treated eyes (31.5 percent) than control eyes (48 percent) that were blind (P<0.001). Of those eyes that had a favorable structural outcome, with or without retinal ablation (cryotherapy to destroy the fringe of the retina through freezing), only a small percentage had best corrected visual acuity better than or equal to 20/40 at age 5 1/2 years (13 percent in the treated group; 17 percent in the untreated control group (P=0.19)). Among the 1398 followed from the 5 large natural history centers of the CRYO-ROP follow-up study, children with retinal residua of ROP (structural changes) had measurable visual acuity that was severly affected and tended to worsen with age. The CRYO-ROP Study proved conclusively that peripheral retinal ablation improves the chances of avoiding blindness, but at least 80 percent of eyes are left with acuity less than 20/40.

Two concerns emerged from the CRYO-ROP extensive study on the natural history of ROP and treatment of threshold ROP. The first of these is failure of peripheral retinal ablation to eliminate all, or nearly all cases, of retinal detachment due to ROP. In the CRYO-ROP Study, 26 percent of eyes with threshold disease in zone II and 78 percent of eyes with zone I threshold disease had an unfavorable structural outcome despite treatment. The second concern is that most children who developed threshold ROP disease had visual acuity worse than 20/40 even if the eye had a favorable structural outcome.

Since no other treatment has yet been shown to be effective in preventing blindness from ROP, retinal ablation remains the treatment of choice. The ETROP Study will test whether earlier treatment is more effective than treatment at threshold in improving functional (visual acuity) outcome following ROP, as well as determining whether earlier treatment decreases the probability of an unfavorable structural outcome.

Earlier treatment is defined as retinal ablation administered to the avascular retina when an eye reaches high risk prethreshold retinopathy of prematurity (ROP). Prethreshold indicates any Zone I ROP; or Zone II stage 2 with plus disease, or stage 3; or Zone II with less than 5 contiguous or 8 cumulative clock hours of stage 3 ROP with plus disease. Recognizing that a substantial number of eyes undergo spontaneous resolution of ROP, eyes will be randomized to early treatment only when high risk for an unfavorable visual acuity outcome is identified. High risk will be determined using a risk model analysis program based on longitudinal natural history data obtained from the CRYO-ROP study. This model integrates risk factors to assign a risk of progression to blindness without treatment. These factors include birth weight, gestational age, ethnicity, singleton/multiple status, outborn status, Zone on first exam, severity of ROP and rate of progression of ROP. When an infant develops prethreshold ROP and greater than or equal to 15 percent risk of unfavorable outcome, randomization to early treatment of one eye will occur. Visual acuity outcome will be measured by masked observers after wearing best correction using the Teller Acuity Card Procedure at 9 months corrected age.

ELIGIBILITY:
Infants <1251 grams birthweight born at participating centers and/or examined by 42 days of life are eligible. The early treatment trial requires that an infant have prethreshold retinopathy of prematurity (ROP).

Ages: 0 Years to 42 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: William V. Good, M.D., Study Chair — Smith-Kettlewell Eye Research Institute
Locations (26):
- United States (26):
  - Stanford University School of Medicine, Palo Alto, California
  - Smith-Kettlewell Eye Research Institute, San Francisco, California
  - UIC Eye Center Department of Ophthalmology and Visual Sciences The Lions of Illinois Eye Research Institute, Chicago, Illinois
  - Indiana University Department of Pediatrics, Indianapolis, Indiana
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - The Zanvyl Krieger Children's Eye Center, Baltimore, Maryland
  - Tufts University School of Medicine Department of Pediatrics, Boston, Massachusetts
  - Pediatric Ophthalmology Associates, PC, Dearborn, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Cardinal Glennon Children's Hospital Neonatology Office, St Louis, Missouri
  - The Children's Hospital of Buffalo Department of Ophthalmology, Buffalo, New York
  - Edward S. Harkness Eye Institute, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Eastern Long Island Retina Associate, Shirley, New York
  - Duke University Eye Center, Durham, North Carolina
  - Columbus Children's Hospital, Columbus, Ohio
  - The Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Oregon Health Sciences University Casey Eye Institute, Portland, Oregon
  - The Children's Hospital of Philadelphia Division of Pediatric Ophthalmology, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine Feigin Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - John Moran Eye Center University of Utah Health Sciences Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Wallace DK, Bremer DL, Good WV, Fellows R, Summers CG, Tung B, Hardy RJ. Correlation of recognition visual acuity with posterior retinal structure in advanced retinopathy of prematurity. Arch Ophthalmol. 2012 Dec;130(12):1512-6. doi: 10.1001/archophthalmol.2012.2118. PMID 22892757
- [Derived] Good WV, Hardy RJ, Wallace DK, Bremer D, Rogers DL, Siatkowski RM, De Becker I, Summers CG, Fellows R, Tung B, Palmer EA. beta-Blocking and racial variation in the severity of retinopathy of prematurity. Arch Ophthalmol. 2012 Jan;130(1):117-8. doi: 10.1001/archopht.130.1.117. No abstract available. PMID 22232483
- [Derived] VanderVeen DK, Bremer DL, Fellows RR, Hardy RJ, Neely DE, Palmer EA, Rogers DL, Tung B, Good WV; Early Treatment for Retinopathy of Prematurity Cooperative Group. Prevalence and course of strabismus through age 6 years in participants of the Early Treatment for Retinopathy of Prematurity randomized trial. J AAPOS. 2011 Dec;15(6):536-40. doi: 10.1016/j.jaapos.2011.07.017. PMID 22153396
- [Derived] Early Treatment for Retinopathy of Prematurity Cooperative Group; Dobson V, Quinn GE, Summers CG, Hardy RJ, Tung B, Good WV. Grating visual acuity results in the early treatment for retinopathy of prematurity study. Arch Ophthalmol. 2011 Jul;129(7):840-6. doi: 10.1001/archophthalmol.2011.143. PMID 21746974
- [Derived] Quinn GE, Dobson V, Hardy RJ, Tung B, Palmer EA, Good WV; Early Treatment for Retinopathy of Prematurity Cooperative Group. Visual field extent at 6 years of age in children who had high-risk prethreshold retinopathy of prematurity. Arch Ophthalmol. 2011 Feb;129(2):127-32. doi: 10.1001/archophthalmol.2010.360. PMID 21320954
- [Derived] Christiansen SP, Dobson V, Quinn GE, Good WV, Tung B, Hardy RJ, Baker JD, Hoffman RO, Reynolds JD, Rychwalski PJ, Shapiro MJ; Early Treatment for Retinopathy of Prematurity Cooperative Group. Progression of type 2 to type 1 retinopathy of prematurity in the Early Treatment for Retinopathy of Prematurity Study. Arch Ophthalmol. 2010 Apr;128(4):461-5. doi: 10.1001/archophthalmol.2010.34. PMID 20385942
- [Derived] Early Treatment for Retinopathy of Prematurity Cooperative Group; Good WV, Hardy RJ, Dobson V, Palmer EA, Phelps DL, Tung B, Redford M. Final visual acuity results in the early treatment for retinopathy of prematurity study. Arch Ophthalmol. 2010 Jun;128(6):663-71. doi: 10.1001/archophthalmol.2010.72. Epub 2010 Apr 12. PMID 20385926